CLINICAL TRIAL: NCT04826718
Title: Associated Factors in the Transmission and Dynamics of SARS-CoV-2 Infection Among Health Care Workers in Hospitals on the Islands of Santiago and São Vicente in Cabo Verde
Brief Title: SARS-CoV-2/COVID-19 Infection Among Health Care Workers
Status: Completed | Type: Observational
Sponsor: Universidade de Cabo Verde (Other)
Collaborators: University of Southern Denmark (Other); Institute of Hygiene and Tropical Medicine, NOVA University, Lisbon, Portugal (Unknown); National Institute of Public Health of Cape Verde, Praia, Cape Verde (Unknown); Centro de Investigacao em Saude de Manhica (Other); European and Developing Countries Clinical Trials Partnership (EDCTP) (Other Government); Bandim Health Project, Bissau, Guinea-Bissau (Unknown)
Responsible Party: Sponsor
Other Study IDs: RIA2020ER-3049
Record Dates: First submitted 2021-03-10; First posted 2021-04-01 (Actual); Last update posted 2023-06-09 (Actual); Status verified 2023-06

CONDITIONS: SARS-CoV-2; BCG; Health Care Worker; COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples Without DNA — Blood.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Cohort: All Health Care Worker (HCW) from Hospital in Santiago and S. Vicente islands, Cabo Verde
- Control: HCW who report no SARS-CoV-2 infection in the period prior to the interview and/or suspected COVID-19 in the period prior to the interview
  Interventions: Other: Questionaire
- Cases: HCW who report positive SARS-CoV-2 infection confirmed by performing a positive PCR test and/or positive Rapid Antigen Test in the period prior to the interview
  Interventions: Other: Questionaire

INTERVENTIONS:
Other: Questionaire — A questionnaire will be administered to all participants to evaluate exposures related to infection at the baseline (enrollement) - Baseline questionnaire. A Follow-up questionnaire to all participants will be done after 3 and 6 months.
  Capillary blood collection, for diagnosis of anti-SARS-CoV-2 Antibodies by rapid test, will be done at the first interview, for all participants (cases and controls).
  Collection of peripheral venous blood, for analysis of the presence and duration of anti-SARS-CoV-2 Antibodies (N and S) will be done at the first interview, and after 6 months for all participants (cases and controls).
  Other Names: SARS-CoV-2 Serology (POC Test); SARS-CoV-2 Serology (ELISA Test)
  Groups: Cases; Control

SUMMARY:
The present study finds opportunities and justifications, taking into consideration that the nature of professional practice in health needs scientific evidence resulting from systematic and systemic studies to strengthen the basis for the decisions made to have an impact on various levels, from the patient to health management itself. In addition, Cabo Verdean authorities may benefit from new evidence obtained by this study. It intends, in a growing number of health professionals exposed or infected with SARS-CoV-2, in the different health structures of the country, to contribute to substantiate a better perception of the problem and the required solutions. Therefore, assessing the potential risk factors for SARS-CoV-2 infection among healthcare workers will be essential to characterize virus transmission, preventing future infections in them and providing the associated healthcare. Due to the advances and important changes described, questions arise that guide this research and allow us to identify the problem.

DETAILED DESCRIPTION:
The problem is stated in the following starting questions:

What conditions and factors are associated with infection and non-infection by SARS-CoV-2 among health professionals working in the three hospitals on the islands of Santiago and São Vicente? Which are they (gender, age group, profession, type of contact, etc.)? Where do the infected HCW typically work (sector)? When and how did the infection occur? What is the prevalence of SARS-CoV-2 antibody in professionals with confirmed SARS-CoV-2 infection and in HCW that thought they were not infected by SARS-CoV-2? How long do anti-SARS-CoV-2 antibodies last? What is the impact of infection on unplanned absenteeism? Which symptoms and complaints (if any) persists after SARS-CoV-2 infection?

ELIGIBILITY:
Inclusion Criteria:

* Being a healthcare professional working in one of the hospitals where the study will take place
* Be aged ≥18 years;
* Cases: SARS-CoV-2 infection confirmed by PCR test and/or Rapid Antigen Test;
* Control: No evidence and/or record of past infection with SARS-CoV-2.

Exclusion Criteria:

* Case: Confirmation of diagnosis test for SARS-CoV-2 without indication of specimen collection date.
* Control: Suspected SARS-CoV-2 infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The population of the study is composed of health professionals working in the Hospitals of the islands of Santiago and S. Vicente.
  In addition to measuring infection-related exposures, specific SARS-CoV-2 infection-related parameters will also be assessed, including presence and duration of anti-SARS-CoV-2 antibodies; absenteeism due to infection; and self-reported symptomatology due to SARS-CoV-2/ COVID-19 infection. All participants be followed up to measure unplanned, infection-related absenteeism, illness-related symptomatology at 3 of for a period of 6 months. At 6 months after enrollement, all participants will also be assessed, including screening of presence of anti-SARS-CoV-2 antibodies (anti-N and anti-S).
Sampling Method: Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2021-09-08 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Total number of days absent from work due to COVID-19 | From March 2020 to March 2022
  Absenteeism due to COVID-19 related symptoms
Unplanned Absenteeism | 6 months after inclusion
  Unplanned absenteeism following SARS-CoV-2 infection
Symptomatology after infection by SARS-CoV-2 | 6 months after inclusion
  If have or not any symptomes after SARS-CoV-2 infection
Presence or absence of anti-SARS-CoV-2 Acs | 6 months after inclusion
  Presence or not of anti-SARS-CoV-2 Anti-N and anti-S
Duration of anti-SARS-CoV-2 Acs | After infection
  Time of duration of anti-SARS-CoV-2 Anti-N and anti-S

CONTACTS AND LOCATIONS:
Overall Officials: Isabel I Araújo, PhD, Principal Investigator — Universidade de Cabo Verde
Locations (1):
- Universidade de Cabo Verde, Praia, Santiago, Cabo Verde

IPD SHARING:
Plan to Share IPD: No